CLINICAL TRIAL: NCT01640782
Title: Open Label, Randomised, Multicenter Phase III Study of Adjuvant Chemotherapy in Radically Resected Adenocarcinoma of the Stomach or Gastroesophageal Junction: Comparison of a Sequential Treatment (CPT-11+5-FU/LV --> TXT+CDDP) Versus a 5-FU/LV Regimen
Brief Title: Intergroup Trial of Adjuvant Chemotherapy in Adenocarcinoma of the Stomach
Acronym: ITACA-S
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other); Gruppo Oncologico Italiano di Ricerca Clinica (Other); Gruppo Oncologico del Nord-Ovest (Other); Italian Trial in Medical Oncology (Other); Southern Italy Cooperative Oncology Group (Other); Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other); Oncotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITACA-S
Record Dates: First submitted 2012-07-09; First posted 2012-07-16 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2013-12

CONDITIONS: Adenocarcinoma of the Stomach; Adenocarcinoma of the Gastroesophageal Junction
Keywords: adenocarcinoma of the stomach; adenocarcinoma of the gastroesophageal junction
MeSH Terms: interventions — Irinotecan; Leucovorin; Fluorouracil; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential regimen (Experimental): Sequential treatment with CPT-11 plus Fluorouracil (FU), folinic acid (LV) and Docetaxel (TXT) plus Cisplatin (CDDP)
  Interventions: Drug: Irinotecan, Leucovorin, 5-Fluorouracil, Docetaxel, Cisplatin
- De Gramont regimen (Active Comparator): Fluorouracil (5-FU), folinic acid (LV)
  Interventions: Drug: Leucovorin, 5-Fluorouracil

INTERVENTIONS:
Drug: Irinotecan, Leucovorin, 5-Fluorouracil, Docetaxel, Cisplatin — * Irinotecan (CPT-11) 180 mg/m2, given as 60 min. i.v. infusion on day 1 every 2 weeks followed by
  * Leucovorin (LV) 100 mg/m2, given as a 2h i.v. infusion on days 1 and 2 every 2 weeks followed by
  * 5-Fluorouracil (5-FU) 400 mg/m2 given as bolus, and then 5-Fluorouracil (5-FU) 600 mg/m2 given as a 22h continuous infusion on days 1 and 2, every 2 weeks for 4 administrations.
  After 3 weeks from last infusion:
  * Docetaxel (TXT) 75 mg/m2, given as a 1h i.v. infusion on day 1 followed by
  * Cisplatin (CDDP) 75 mg/m2, given as a 1h i.v. infusion on.day 1, every 3 weeks, for 3 cycles.
  Arms: Sequential regimen
Drug: Leucovorin, 5-Fluorouracil — * Leucovorin (LV) 100 mg/m2, given as a 2h i.v. infusion on days 1 and 2 every 2 weeks followed by
  * 5-Fluorouracil (5-FU) 400 mg/m2 given as bolus, and then 5-Fluorouracil (5-FU) 600 mg/m2 given as a 22h continuous infusion on days 1 and 2, every 2 weeks for 9 administrations.
  Arms: De Gramont regimen

SUMMARY:
Open label, randomised, multicenter, superiority study for efficacy. Patients with histologically proven adenocarcinoma of the stomach or gastroesophageal junction without gross or microscopic evidence of residual disease after surgery with curative intent and fulfilling all the inclusion/exclusion criteria are eligible for this study.

DETAILED DESCRIPTION:
Open label, randomised, multicenter, superiority study for efficacy. Patients with histologically proven adenocarcinoma of the stomach or gastroesophageal junction without gross or microscopic evidence of residual disease after surgery with curative intent and fulfilling all the inclusion/exclusion criteria are eligible for this study.

Allocation to treatment will be done centrally using a randomisation scheme and will be stratified by center and nodal involvement (N- vs. N+). Access to random system will be allowed by phone or via web.

All included patients in both groups will received fixed period of 18 weeks of treatment unless unacceptable toxicity or disease relapse during treatment. After cessation of therapy, patients will have a follow-up period while not receiving further treatment. After relapse further chemotherapy is left to the investigator's judgement. When the last patient is randomised, follow-up will be truncated at the achievement of the required number of events.

Time to progression and time to death are the main study outcomes. During the course of the trial, an independent Data and Safety Monitoring Board (DSMB) will advise the Steering Committee on efficacy and/or safety aspects of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach or gastroesophageal junction without gross or microscopic evidence of residual disease after surgery with curative intent;
* Subtotal or total gastrectomy with at least D1 dissection;
* Gastroesophageal junction adenocarcinoma extending to the stomach with the center lying 2 to 5 cm below the anatomic esophago-gastric junction;
* Patients with nodal involvement (pN+) or patients without nodal involvement (pN0) with pT2b-3-4. It is recommended to examine at least 15 lymph nodes;
* Age between 18 and 75 years;
* ECOG performance status 0-1;
* No previous chemotherapy and/or radiotherapy;
* Complete staging procedures within 3 months prior to randomization;
* Laboratory requirement (within 8 days prior to randomization):

  * Haematology (Neutrophils > 2.0 x 109 /L, Platelet > 100 x 109 /L, Hemoglobin > 10g/dL);
  * Hepatic function (Total bilirubin < 1 UNL, ASAT (SGOT) and ALAT (SGPT) < 2.5xUNL, Alkaline phosphatase < 2.5xUNL. Patients with ASAT or ALAT > 1.5xUNL associated with alkaline phosphatase > 2.5XUNL are not eligible.)
  * Renal function (Creatinine < 1.5 UNL. In presence of borderline values, the calculated creatinine clearance according to Cockroft-Gault formula, 60 ML/min.
* Recovery from acute effects of surgery. The first infusion of study chemotherapy should be administered 3 to 8 weeks after surgery treatment;
* Written informed consent signed and dated before randomization procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirement.

Exclusion Criteria:

* Non-radical surgery as assessed microscopically (no tumor-free margin of resection, positive biopsy of peritoneal suspicious lesions);
* Synchronous metastases, even curatively resected;
* Pregnant or lactating patients; patients with reproductive potential must implement adequate contraceptive measures;
* Prior or concurrent history of:

  * positive HIV serology,
  * chronic diarrhoea,
  * chronic bowel inflammation or subobstruction,
  * neoplasm other than gastric cancer, except for: curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix,
  * previous history of myocardial infarction within 1 year from study entry,
  * hypersensitivity reaction to polysorbate 80;
* Presence of other systemic disease limiting drug administration and influencing patient survival:

  * uncontrolled hypertension,
  * high-risk uncontrolled arrhythmia,
  * unstable angina pectoris;
* Symptomatic

  * peripheral neuropathy,
  * altered hearing > 2 grade by NCIC-CTG criteria;
* Active uncontrolled infection.
* Definite contra-indications for the use of corticosteroids: unstable diabetes mellitus, active peptic ulcer;
* Concurrent administration of:

  * corticosteroids or equivalent except as use for the prophylactic medication regimen, treatment of acute hypersensitivity reactions or unless chronic treatment (initiated > 6 months prior to study entry) at low doses (< 20mg methylprednisolone or equivalent);
  * any other experimental drug under investigation: concurrent treatment with any other anticancer therapy, growth factors with preventive intent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2005-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival will be defined as the time from date of randomisation to date of first appearance of local, regional or distant relapse, or death from any cause; patients alive without relapse will be censored at date last known to be alive. | 3 years

SECONDARY OUTCOMES:
OS will be defined as the time from date of randomisation to date of death by any cause, with living patients censored at date last known to be alive | 3 years
Toxicity, graded according to the NCI-CTG Expanded Common Toxicity Criteria | 3 years
Adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Bajetta, MD, Principal Investigator — Istituto Nazionale Per lo Studio e la Cura dei Tumori Milano
Locations (101):
- Italy (101):
  - ASL 6 - Fabriano, Fabriano, Ancona
  - Ospedale Civile di Senigallia, Senigallia, Ancona
  - dell'Azienda Ospedaliero-Universitaria Ospedali Riuniti Umberto I, Torrette Di Ancona, Ancona
  - Ospedale. S. Donato, Arezzo, Arezzo
  - Presidio Ospedaliero di Ariano Irpino, Ariano Irpino, Avellino
  - A.O. "G. Rummo", Benevento, Benevento
  - Ospedali "Riuniti", Bergamo, Bergamo
  - A.O. "Ospedale Treviglio-Caravaggio", Treviglio, Bergamo
  - Ospedale degli Infermi di Biella, Biella, Biella
  - Ospedale Maggiore-Bellaria, Bologna, Bologna
  - A.O.Policlinico "S.Orsola-Malpighi", Bologna, Bologna
  - Ospedale Sant'Orsola - Fatebenefratelli, Brescia, Brescia
  - Casa di Cura Poliambulanza di Brescia, Brescia, Brescia
  - Spedali Civili, Brescia, Brescia
  - P.O. di Monserrato - Policlinico Universitario di Cagliari, Monserrato, Cagliari
  - P.O. di Monserrato, Monserrato, Cagliari
  - P.O. Vittorio Emanuele, Catania, Catania
  - Ospedale Garibaldi in Nesima, Catania, Catania
  - A.O. Sant'Anna, Como, Como
  - Ospedale "Valduce", Como, Como
  - Ospedale Civile "Ferrari", Castrovillari, Cosenza
  - Presidio Ospedaliero di Lamezia Terme, Lamezia Terme, Cosenza
  - Ospedale "San Francesco" di Paola, Paola, Cosenza
  - A.O. "Ospedale Maggiore" di Crema, Crema, Crema
  - Azienda Ospedaliera "Istituti Ospitalieri" di Cremona, Cremona, Cremona
  - P.O. S. Lazzaro, Alba, Cuneo
  - A.O. "S.Croce e Carle", Cuneo, Cuneo
  - Azienda Ospedaliera Universitaria "S.Anna", Ferrara, Ferrara
  - Ospedale Santa Maria Annunziata, Antella, Firenze
  - Ospedale "San Giuseppe", Empoli, Firenze
  - A.O. Universitaria Careggi, Florence, Firenze
  - A.O. "G.B.Morgagni-L.Pierantoni, Forlì, Forli
  - E.O. Ospedali Galliera di Genova, Genova, Genova
  - Istituto Nazionale per la Ricerca sul Cancro, Genova, Genova
  - P.O. "A.Manzoni" di Lecco, Lecco, Lecco
  - Azienda USL 6 - P.O. Livorno, Livorno, Livorno
  - Ospedale Civile di Casalpusterlengo, Lodi, Lodi
  - Ospedale "Campo di Marte", Lucca, Lucca
  - A.O. "C.Poma", Mantova, Mantova
  - Ospedale Civico di Carrara, Carrara, Massa Carrara
  - Istituto Scientifico Universitario San Raffaele, Milan, Milano
  - Istituto Nazionale per la cura dei tumori, Milan, Milano
  - Istituto Europeo di Oncologia, Milan, Milano
  - Azienda Ospedaliera "Ospedale San Carlo Borromeo", Milan, Milano
  - Azienda Ospedaliera "Luigi Sacco" Polo Universitario, Milan, Milano
  - Azienda Ospedaliera "San Paolo" Polo Universitario, Milan, Milano
  - A.O "San Gerardo" di Monza, Monza, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Ospedale IRCCS Policlinico di San Donato, San Donato Milanese, Milano
  - Presidio Ospedaliero "Serbelloni"di Gorgonzola, Vizzolo Predabissi, Milano
  - Ospedale "B.Ramazzini", Carpi, Modena
  - A.O. "D.Cotugno", Napoli, Napoli
  - A.O.R.N. "Antonio Cardarelli", Napoli, Napoli
  - Azienda Ospedaliera Universitaria "Federico II", Napoli, Napoli
  - Istituto Nazionale per lo Studio e la Cura dei Tumori "Fondazione Pascale", Napoli, Napoli
  - Presidio Ospedaliero "Santa Maria delle Grazie", Pozzuoli, Napoli
  - Azienda Ospedaliera "Maggiore della Carità", Novara, Novara
  - Ospedale Civile di Este, Este, Padova
  - Azienda Ospedaliera di Padova, Padua, Padova
  - Ospedali "Civico e Benfratelli - G. Di Cristina - Maurizio Ascoli", Palermo, Palermo
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone"di Palermo, Palermo, Palermo
  - Azienda Ospedaliera di Parma, Parma, Parma
  - Ospedale di Città di Castello - ASL 1 Umbria, Città di Castello, Perugia
  - Ospedale di Marsciano - Servizio Oncologico, Marsciano, Perugia
  - Ospedale "Santa Croce", Fano, Pesaro
  - Ospedale Civile "San Massimo", Penne, Pesaro
  - A.O."Ospedale S.Salvatore", Pesaro, Pesaro
  - Ospedale Civile dello "Spirito Santo", Pescara, Pescara
  - Ospedale Civile di Piacenza, Piacenza, Piacenza
  - Azienda Ospedaliera-Universitaria Pisana, Pisa, Pisa
  - Centro di Riferimento Oncologico - INT, Aviano, Pordenone
  - A.O. "Santa Maria degli Angeli", Pordenone, Pordenone
  - Ospedale "San Carlo"di Potenza, Potenza, Potenza
  - Centro di Riferimento Oncologico di Basilicata, Rionero in Vulture, Potenza
  - Ospedale "Misericordia e Dolce", Prato, Prato
  - P.O. di Faenza, Faenza, Ravenna
  - P.O. Umberto I di Lugo, Lugo, Ravenna
  - P.O. di Ravenna - Azienda Unità Sanitaria Locale di Ravenna, Ravenna, Ravenna
  - A.O. "Bianchi-Melacrino-Morelli", Reggio Calabria, Reggio Calabria
  - Ospedale Civile di Siderno, Siderno, Reggio Calabria
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Reggio Emilia
  - Ospedale "Infermi", Rimini, Rimini
  - Azienda Ospedaliera Universitaria "Policlinico Tor Vergata", Roma, Roma
  - Policlinico Umberto I, Roma, Roma
  - Ospedale Fatebenefratelli "San Giovanni Calibita", Roma, Roma
  - Istituto Nazionale di Riposo e Cura per Anziani, Roma, Roma
  - Istituto Dermopatico dell'Immacolata - IRCCS, Roma, Roma
  - Ospedale "San Luca", Vallo della Lucania, Salerno
  - Azienda Unità Sanitaria Locale n°1 Sassari, Sassari, Sassari
  - Ospedale Civile di Sassari, Sassari, Sassari
  - A.O. della Valtellina e della Valchiavenna, Sondrio, Sondrio
  - Istituto per la Ricerca e la Cura del Cancro di Candiolo, Candiolo, Torino
  - Ospedale San Giovanni Battista di Torino, Torino, Torino
  - Ospedale Civile di Latisana, Latisana, Udine
  - Azienda Ospedaliera S. Maria, Terni, Umbria
  - Presidio Ospedaliero di Saronno - A.O. "Ospedale di Circolo di Busto Arsizio", Saronno, Varallo
  - A.O. "Ospedale di Circolo di Busto Arsizio", Busto Arsizio, Varese
  - A.O."Ospedale di Circolo e Fondazione Macchi", Varese, Varese
  - Ospedale di Legnago, Legnago, Verona
  - A.O. Istituti Ospitalieri di Verona, Verona, Verona
  - Ospedale di Montecchio Maggiore, Montecchio Maggiore, Vicenza

REFERENCES:
- [Derived] Bajetta E, Floriani I, Di Bartolomeo M, Labianca R, Falcone A, Di Costanzo F, Comella G, Amadori D, Pinto C, Carlomagno C, Nitti D, Daniele B, Mini E, Poli D, Santoro A, Mosconi S, Casaretti R, Boni C, Pinotti G, Bidoli P, Landi L, Rosati G, Ravaioli A, Cantore M, Di Fabio F, Aitini E, Marchet A; ITACA-S (Intergroup Trial of Adjuvant Chemotherapy in Adenocarcinoma of the Stomach Trial) Study Group. Randomized trial on adjuvant treatment with FOLFIRI followed by docetaxel and cisplatin versus 5-fluorouracil and folinic acid for radically resected gastric cancer. Ann Oncol. 2014 Jul;25(7):1373-1378. doi: 10.1093/annonc/mdu146. Epub 2014 Apr 12. PMID 24728035